CLINICAL TRIAL: NCT04065191
Title: High-intensity Interval Training for Workplace Health Promotion: Evaluation of Feasibility and Preventive Effects in a Real-World Setting
Brief Title: Workplace HIIT: Feasibility and Preventive Effects of HIIT in the Real-World
Acronym: WORK-HIIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WORK-HIIT-Study
Record Dates: First submitted 2019-05-15; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Primary Prevention; Health Promotion
Keywords: Aerobic exercise; Cardiorespiratory Fitness; High-intensity interval training (HIIT); Workability; Prevention
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-intensity interval training (Experimental): High-intensity interval training
  Interventions: Other: High-intensity interval training

INTERVENTIONS:
Other: High-intensity interval training — Heart rate based high-intensity interval training

SUMMARY:
The aim of this study is to investigate the effects of an extremely time-efficient high-intensity interval training program, performed over a period of six months in a real-world (workplace) setting, on cardiorespiratory fitness, cardiometabolic risk profile, and self-reported outcomes including perceived stress and subjective work ability in previously sedentary employees.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary Lifestyle over at least 1 year prior to the study

Exclusion Criteria:

* Pregnancy, Lactation
* Psychological disorders, epilepsy, sever neurological disorders
* Participation in other exercise- or nutrition studies within the last 6 months
* coronary heart disease, heart failure
* malignant disease
* severe rheumatic or neurological disease
* severe/unstable hypertension (resting RR: >180/>110 mmHg)
* severely restricted lung function (FEV1 <60%)
* unstable Diabetes mellitus
* severe orthopedic disease/restriction
* acute / chronic infectious diseases
* Electronic implants (defibrillator, pacemaker)
* Persons in mental hospitals by order of authorities or jurisdiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness (CRF) | 12 months [Change from Baseline to 6 months and Change from Baseline to 6 months after the end of the intervention]
  CRF will be assessed by measuring maximum oxygen uptake (VO2max)

SECONDARY OUTCOMES:
Metabolic Syndrome Z-Score (MetS-Z-Score) | 12 months [Change from Baseline to 6 months and Change from Baseline to 6 months after the end of the intervention]
  MetS-Z-Score will be calculated from each individual's measures of waist circumference (cm), mean arterial blood pressure (mmHg), Glucose (mg/dL), triglycerides (mg/dL), and HDL-cholesterol (mg/dL), based on equations specific to sex.
Muscle mass | 12 months [Change from Baseline to 6 months and Change from baseline to 6 months after the end of the intervention]
  Muscle mass (kg) will be measured by Bioelectrical Impedance Analysis (BIA)
Fat mass | 12 months [Change from baseline to 6 months and change from baseline to 6 months after the end of the intervention]
  Fat mass (kg) will be measured by Bioelectrical Impedance Analysis (BIA)
Total body water | 12 months [Change from baseline to 6 months and change from baseline to 6 months after the end of the intervention]
  Total body water (l) will be measured by Bioelectrical Impedance Analysis (BIA)
Insulin sensitivity | 12 months [Change from Baseline to 6 months and Change from Baseline to 6 months after the end of the intervention]
  Insulin sensitivity will be estimated using homeostasis model assessment index (HOMA)
Inflammation status | 12 months [Change from Baseline to 6 months and Change from Baseline to 6 months after the end of the intervention]
  Inflammation status will be assessed by measuring blood levels (mg/L) of c-reactive protein (CRP) and high-sensitivity c-reactive protein (hs-CRP)
Health-related quality of life | 12 months [Change from Baseline to 6 months and Change from Baseline to 6 months after the end of the intervention]
  Health-related quality of life will be assessed by using the standardized and validated EQ-5D-5L Questionnaire, consisting of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient ticks the box next to the most appropriate statement in each dimension (scale: 1-5; lower value = better outcome). The digits for the 5 dimensions can be combined into a 5-digit number that describes the patient's health state.The EQ VAS records the patient's self-rated health on a vertical visual analogue scale (0-100, higher value = better outcome).
Pain scores | 12 months [Change from Baseline to 6 months and Change from Baseline to 6 months after the end of the intervention]
  Pain scores will be assessed by using the standardized and validated Chronic Pain Grade Questionnaire (CPGQ). The CPGQ is a seven-item instrument to evaluate overall severity of chronic pain based on 2 dimensions: pain intensity and pain-related disability. The responses on the 7 items are used to compute scores for 3 subscales: pain intensity (0-100), disability score (0-3), and disability Points (0-3). Lower values indicate better outcomes.
  moderately limiting intensity (Grade III), high disability and severely limiting intensity (Grade IV) (see Von Korff et al 1992).
Perceived stress | 12 months [Change from Baseline to 6 months and Change from Baseline to 6 months after the end of the intervention]
  Perceived stress will be assessed by using the standardized and validated Perceived Stress Questionnaire (PSQ). The PSQ comprises different components of stress (worries, tension, joy, demands), with 5 items each. It contains both positively and negatively formulated items in order to reduce acquiescent bias. Each item is answered using a four-point Likert-type scale, ranging from 1 to 4. Higher scores indicate more severe perceived stress.
Subjective work ability | 12 months [Change from Baseline to 6 months and Change from Baseline to 6 months after the end of the intervention]
  Subjective work ability will be assessed by using the standardized and validated Work Ability Index Questionnaire (WAI). WAI obtains information related to diseases, functional limitations, sick leave, and mental resources. The questionnaire consistes of 7 items, including current work ability compared with the lifetime best (item 1, 0-10), work ability in relation to the demands of the job (item 2, 2-10), number of current disease groups diagnosed by a physician (item 3, 1-7), estimated work impairment due to diseases (item 4, 1-6), sick leave during the past year (item 5, 1-5), personal prognosis of work ability for 2 years from now (item 6, 1,4 or 7) and mental resources, referring to the workers life in general, both at work and during leisure time(item 7, 1-4). The total WAI score is calculated by summing up the scores of all items and is ranged from 7 to 49. The total WAI scores are categorized into 4 levels: poor (7-27), moderate (28-36), good (37-43), and excellent (44-49).

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Reljic, Dr., Principal Investigator — University Erlangen Nuremberg Medical School; Yurdaguel Zopf, Prof., Principal Investigator — University Erlangen Nuremberg Medical School
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany